CLINICAL TRIAL: NCT03967132
Title: Growth and Tolerance of Young Infants Fed Milk-Based Infant Formula With Oligosaccharides
Brief Title: Growth and Tolerance of Infants Fed Milk-Based Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AL29A
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Gastro-Intestinal Tolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Infant Formula (Active Comparator): Milk-based infant formula
  Interventions: Other: Control Infant Formula
- Experimental Infant Formula (Experimental): Milk-based Infant Formula with oligosaccharides
  Interventions: Other: Experimental Infant Formula
- Reference Group (Other): Human-milk fed
  Interventions: Other: Reference Group

INTERVENTIONS:
Other: Control Infant Formula — Ready to feed infant formula, feed ad libitum
  Arms: Control Infant Formula
Other: Experimental Infant Formula — Ready to feed infant formula, feed ad libitum
  Arms: Experimental Infant Formula
Other: Reference Group — Human milk, breast feeding ad libitum
  Arms: Reference Group

SUMMARY:
The purpose of this study is to evaluate growth and tolerance of healthy term infants fed an experimental milk-based infant formula with oligosaccharides compared to a control milk-based infant formula.

ELIGIBILITY:
Inclusion Criteria:

* Good health as determined from participant's medical history
* Singleton from a full-term birth with a gestational age of 37-42 weeks
* Birth weight was > 2490 g (~5 lbs. 8 oz.)
* If parent(s) of the participant elect to formula-feed the participant, parent(s) confirm the participant has not been given human milk since being discharged from the hospital following birth, and confirm their intention to feed their infant the study product as the sole source of feeding from Study Visit 1-Visit 7, unless instructed otherwise by their healthcare professional.
* If parent(s) of the participant elect to feed the infant human milk, they confirm the infant has not received any formula prior to enrollment, and confirm their intention to exclusively feed human milk from birth, and as the sole source of feeding from Study Visit 1-Visit 7.
* Parent(s) confirm their intention not to administer vitamin or mineral supplements (with the exception of Vitamin D supplements), solid foods or juices to their infant from enrollment through the duration of the study, unless instructed otherwise by their healthcare professional.
* Participant's parent(s) has voluntarily signed and dated an ICF, approved by an IRB/IEC and provided HIPAA (or other applicable privacy regulation) authorization prior to any participation in the study.

Exclusion Criteria:

* An adverse maternal, fetal or participant medical history that is thought by the investigator to have potential for effects on tolerance, growth, and/or development.
* Participant is taking and plans to continue taking medications (including over the counter (OTC), such as Mylicon® for gas), prebiotics, probiotics, home remedies (such as juice for constipation), herbal preparations or rehydration fluids that might affect GI tolerance.
* Participant participates in another study that has not been approved as a concomitant study by AN.

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 189 (Actual)
Dates: Start 2019-06-08 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Weight | Day of life 14 - 119
  Weight gain per day

SECONDARY OUTCOMES:
Stool Characteristics | Study Day 1 to Day of life 119
  Parent completed diary
Formula Tolerance | Study Day 1 to Day of life 119
  Parent completed diary
Length | Study Day 1 to Day of life 119
  Length gain per day
Head Circumference (HC) | Study Day 1 to Day of life 119
  HC gain per day
Illness Incidence | Study Day 1 to Day of life 119
  Parent reported incidence of illness

OTHER OUTCOMES:
Stool Sample | Study Day 1 to Day of life 119
  Microbiota characterization

CONTACTS AND LOCATIONS:
Overall Officials: Timberly Williams, PhD, Study Chair — Abbott Nutrition
Locations (19):
- United States (19):
  - Watching Over Mothers & Babies, Tucson, Arizona
  - Pediatric Medical Associates, Sacramento, California
  - Norwich Pediatric Group, P.C., Norwich, Connecticut
  - Phoenix Medical Research LLC, Miami, Florida
  - University Clinical Research-Deland, LLC a/b/a Accel Clinical Research, Orlando, Florida
  - Clinical Research Prime, Idaho Falls, Idaho
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Michael W. Simon, M.D., PSC, Nicholasville, Kentucky
  - Springs Medical Research, Owensboro, Kentucky
  - Institute of Clinical Research, LLC, Mentor, Ohio
  - The Cleveland Pediatric Research Center, LLC, Middleburg Heights, Ohio
  - Holston Medical Group, Kingsport, Tennessee
  - Midsouth Center for Clinical Research, Memphis, Tennessee
  - ARC Clinical Research at Wilson Parke, Austin, Texas
  - Ventavia Research Group, LLC, Fort Worth, Texas
  - Ventavia Research Group, Houston, Texas
  - Ventavia Research Group, LLC 3078, Keller, Texas
  - Kagan Pediatrics - HD Research Corporation, Pearland, Texas
  - Plano Pediatrics - ACRC Trials, Plano, Texas

IPD SHARING:
Plan to Share IPD: No